CLINICAL TRIAL: NCT03223584
Title: Exploratory Study to Inventory Opportunities to Optimize Continuity of Pharmacotherapy at Hospital Discharge
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Joke Wuyts, PharmD, KU Leuven
Other Study IDs: S58480
Record Dates: First submitted 2016-01-25; First posted 2017-07-21 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Pharmacist; Physicians, Primary Care; Patient Discharge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Pharmacists-Leuven: Individual interviews with approximately 5 pharmacists
- Pharmacists-Bruges: Individual interviews with approximately 5 pharmacists
- Pharmacists-Mortsel: A focus group with pharmacists and general practitioners
- General Practitioners-Leuven: Individual interviews with approximately 5 general practitioners
- General Practitioners-Bruges: Individual interviews with approximately 5 general practitioners
- General Practitioners-Mortsel: A focus group with pharmacists and general practitioners

SUMMARY:
Title of the research:

Exploratory study to inventory opportunities to optimize continuity of pharmacotherapy at hospital discharge

Study area:

Care region Leuven (individual interviews), care region Bruges (individual interviews) and care region Mortsel (One focus group).

Aims:

From an explorative angle, the study aims to identify hurdles, barriers, facilitators and needs that general practitioners and community pharmacists experience with patients who have recently been discharged from a hospital. From a feasibility standpoint, the study aims to investigate what supportive actions are feasible and useful to optimize the care process upon hospital discharge. For this purpose, a discharge document for the community pharmacist will be shown to the healthcare professionals. The HCP will be given the opportunity to give feedback on this document.

Study design:

A non-interventional, qualitative study is set up using face-to-face, semi-structured interviews and a focus group.

Study population:

Community pharmacists and general practitioners that are employed in the study region and that are considered opinion leaders.

Number of health care professionals:

Individual interviews will be organised until there is saturation of information and no new elements are provided in the interviews. At least five community pharmacists and five general practitioners will be interviewed per care region. In addition, a focus group will take place in care region Mortsel.

Procedures:

Upon an informed consent of the healthcare professional, a semi-structured face-to-face interview will take place. The interview will focus on concrete patient cases, provided by the healthcare professional, as well as a fictional case of the researcher. In the focus group, data of the individual interviews will be presented and the relevance and completeness of the information will be assessed. Finally, the aim of the focus group is to reach a consensus on the research questions.

ELIGIBILITY:
Inclusion Criteria:

* Profession: general practitioner or community pharmacists
* Employment in care regions Leuven, Bruges or Kontich
* Experience in daily practice
* Interest in research or optimisation of the healthcare profession. For example supervisors of an internship, local coordinators of general practitioners or pharmacy clusters and active HCP that are linked with professional associations.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community pharmacists and general practitioners that are employed in the study region and that are considered opinion leaders.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Semi-structured interviews/focus group: Experienced problems and solutions | Approximately 1 hour
  Experienced problems during counseling of discharged older patients and potential solutions
Semi-structured interviews: Strengths and weaknesses of a proposal for a discharge document for community pharmacist (using open ended questions) | Approximately 1 hour
  During the interviews, a proposal for a discharge document will be shown to healthcare professionals. They will be asked to give their feedback on the content of the document (not applicable for the focus group)

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wuyts J, Vande Ginste M, De Lepeleire J, Foulon V. Discharge report for the community pharmacist: Development and validation of a prototype. Res Social Adm Pharm. 2020 Feb;16(2):168-177. doi: 10.1016/j.sapharm.2019.04.049. Epub 2019 Apr 25. PMID 31078447